CLINICAL TRIAL: NCT06075563
Title: Total Lymphoid Irradiation as Conditioning for Pediatric Haploidentical Hematopoietic Stem Cell Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Children's Hospital (Other)
Collaborators: The University of Hong Kong (Other); Hong Kong Sanatorium & Hospital (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAED-2023-020
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-03

CONDITIONS: Hematopoietic Organs; Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Total lymphoid irradiation (TLI)
  Interventions: Radiation: Total lymphoid irradiation

INTERVENTIONS:
Radiation: Total lymphoid irradiation — Total lymphoid irradiation (TLI) 6Gy by tomotherapy as part of conditioning treatment before haploidentical hematopoietic stem cell transplant

SUMMARY:
In this comparative study, the investigators aim to compare prospective pediatric patients who receive total lymphoid irradiation (TLI) using tomotherapy with age- and disease-matched controls who receive conventional total body irradiation (TBI) as part of conditioning for haploidentical hematopoietic stem cell transplantation (HSCT) for both malignant and non-malignant diseases. The investigators shall evaluate graft failure-free, graft-versus-host disease (GVHD)-free survival, overall survival, frequency of rejection, GVHD, relapse of malignancy, adverse effects and post-transplant immunoreconstitution.

DETAILED DESCRIPTION:
Radiotherapy at a dose of 6Gy divided into 3 equal fractions (2Gy per fraction) to all lymphoid organs (TLI) over 2 days using tomotherapy will be given to participants as part of the conditioning treatment before haploidentical hematopoietic stem cell transplantation (HSCT). Retrospective patients who are age- and disease-matched with the recruited patients and had received radiotherapy to the whole body (TBI) with or without lung shielding at a total dose of 2-12 Gy delivered as 1-6 equal fractions by conventional opposed fields radiotherapy as part of conditioning will be compared for the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 0-18 years who requires allogeneic HSCT, has no human leukocyte antigen (HLA)-matched sibling donor but has an HLA-haploidentical donor.
* Adequate organ function to tolerate the conditioning chemotherapy and radiotherapy
* Karnofsky or Lansky performance status score ≥50

Exclusion Criteria:

* Pregnant or lactating woman
* HIV infection
* Patients for whom alternative treatment is deemed more appropriate by treating physician
* Patients who are unlikely to benefit from haploidentical hematopoietic stem cell transplantation, e.g., terminal malignancy with multiorgan failure

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Graft failure-free, GVHD-free survival | up to 1 year
  From the date of treatment start until the date of graft failure or GVHD or death from any cause, whichever comes first, assessed up to 1 year

SECONDARY OUTCOMES:
Overall survival | up to 1 year
  From the date of treatment start until the date of death from any cause, whichever comes first, assessed up to 1 year
Proportion of patients who develop relapse among those with malignant diseases | up to 1 year
  Relapse is defined as reappearance of biopsy-proven malignant disease after complete remission
Proportion of patients who develop graft failure | up to 1 year
  Graft failure is defined as donor cells <5% in whole blood
Proportion of patients who develop acute graft-versus-host disease | up to 1 year
  Acute graft-versus-host disease is defined by MAGIC criteria
Proportion of patients who develop chronic graft-versus-host disease | up to 1 year
  Chronic graft-versus-host disease is defined by NIH criteria
Proportion of patients who develop adverse events not mentioned in outcomes 4-6 | up to 1 year
  Adverse events are graded according to Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events version 5 (CTCAEv5)
Blood T lymphocyte count at 3 months | at 3 months
  Mean T lymphocyte count in blood among evaluable patients
Blood T lymphocyte count at 1 year | at 1 year
  Mean T lymphocyte count in blood among evaluable patients

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cheuk, Principal Investigator — Hong Kong Children's Hospital
Locations (1):
- Hong Kong Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No